CLINICAL TRIAL: NCT01211769
Title: Alcohol Dependence: Study of the Possible Reduction of Compulsion by Association of Naltrexone With Poly-unsaturated Fatty Acids (PUFAs)
Brief Title: Effects of Omegas 3 and 6 on Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Responsible Party: José Carlos Fernandes Galduróz, Adjuncto Professor of UNIFESP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006/01641-6
Record Dates: First submitted 2008-12-05; First posted 2010-09-29 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Alcohol Dependence
Keywords: PUFAs; Alcoholism; Treatment; Effectiveness
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PUFAs (Experimental): Polyunsaturated fatty acids (PUFAs): borage Oil (Borago officinalis L. Boraginaceae) - rich in omega 6 PUFA, dosage of 1 gram; along with 1 gram of fish oil - rich in omega 3 PUFA;
  Interventions: Drug: PUFAs
- Naltrexone (Active Comparator): Naltrexone chlorhydrate 50 mg
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Naltrexone Placebo: pill with 50mg of talcum powder, identical to the pill of naltrexone;
  Polyunsaturated fatty acids Placebo (PUFAs Placebo): yellow liquid paraffin identical to the pills of borage seed and fish oil.
  Interventions: Drug: Placebo
- Naltrexone + PUFAs (Other): Polyunsaturated fatty acids (PUFAs): borage Oil (Borago officinalis L. Boraginaceae) - rich in omega 6 PUFA, dosage of 1 gram; along with 1 gram of fish oil - rich in omega 3 PUFA;
  Naltrexone chlorhydrate 50 mg
  Interventions: Drug: Naltrexone + Placebo

INTERVENTIONS:
Drug: Naltrexone — A pill of naltrexone chlorhydrate 50mg, associated to yellow liquid paraffin pills simulating borage seed and fish oil.
  Arms: Naltrexone
Drug: PUFAs — Borage Oil (Borago officinalis L. Boraginaceae) - rich in omega 6 PUFA, dosage of 1 gram and Fish oil 1 gram - rich in omega 3 PUFAs; associated to a pill with 50mg of talcum powder, identical to the pill of naltrexone.
  Arms: PUFAs
Drug: Placebo — A pill with 50mg of talcum powder, identical to the pill of naltrexone; associated to PUFAs Placebo pills (yellow liquid paraffin identical to the pills of borage seed and fish oil).
  Arms: Placebo
Drug: Naltrexone + Placebo — A pill of naltrexone chlorhydrate 50mg, associated to Borage Oil (Borago officinalis L. Boraginaceae) - rich in omega 6 PUFA, dosage of 1 gram and Fish oil 1 gram - rich in omega 3 PUFAs.
  Arms: Naltrexone + PUFAs

SUMMARY:
Context: The treatment of alcoholism is a challenge for psychiatrists and patients. Some studies have shown that alcohol alters the environment of the membranes, mainly by modifying their permeability through the lipid fraction. These lipids are known as essential fatty acids (EFA) because they are obtained only through the diet, as the human body is unable to synthesize them. Linolenic acid (LA), or omega 6, and alpha-linolenic acid (ALA), or omega 3, are polyunsaturated fatty acids (PUFAs). Finally, ethanol changes the absorption and metabolism of PUFAs, and it's supplementation may be helpful for alcohol dependence recovery.

Objective: to assess the effectiveness of PUFAs supplementation in the treatment of alcohol dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* severe alcohol dependence
* no history of allergic processes, hepatic, cardiovascular, renal, pulmonary, endocrine or neurological pathologies, as well as no history of psychiatric disorders, dependences other than alcohol and/or tobacco, and blood test results outside the reference range

Exclusion Criteria:

* history of allergic processes, hepatic, cardiovascular, renal, pulmonary, endocrine or neurological pathologies
* dependences other than alcohol and/or tobacco
* psychiatric disorders
* test laboratories results outside the reference range

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos F Galduróz, Ph.D, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Fogaca MN, Santos-Galduroz RF, Eserian JK, Galduroz JC. The effects of polyunsaturated fatty acids in alcohol dependence treatment--a double-blind, placebo-controlled pilot study. BMC Clin Pharmacol. 2011 Jul 26;11:10. doi: 10.1186/1472-6904-11-10. PMID 21787433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We comprised the sample through advertisement in newspaper and referral from outpatient services specialized in alcohol dependence treatment. The requirement for their participation was that they were not following any other treatment during the study.
Pre-assignment Details: 645 individuals contacted; 325 were excluded after answering the questionnaire by phone. Most of the remaining 320 patients did not meet the inclusion criteria.
  80 patients participated in the study.
Groups:
- Naltrexone: Naltrexone chlorhydrate 50 mg
  Polyunsaturated fatty acids Placebo (PUFAs Placebo): yellow liquid paraffin identical to the pills of borage seed and fish oil.
- PUFAs: Polyunsaturated fatty acids (PUFAs): borage Oil (Borago officinalis L. Boraginaceae) - rich in omega 6 PUFA, dosage of 1 gram; along with 1 gram of fish oil - rich in omega 3 PUFA;
  Naltrexone Placebo: pill with 50mg of talcum powder, identical to the pill of naltrexone;
Period: Overall Study
Arm/Group | Placebo | Naltrexone | PUFAs | Naltrexone + PUFAs
Started | 20 | 20 | 20 | 20
Participants/Group | 20 | 20 | 20 | 20
Completed | 11 | 10 | 12 | 9
Not Completed | 9 | 10 | 8 | 11
Not completed — Lost to Follow-up | 7 | 9 | 5 | 9
Not completed — Physician Decision | 2 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naltrexone | PUFAs | Naltrexone + PUFAs | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 00 | 00 | 00 | 00 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 80
  >=65 years | 00 | 00 | 00 | 00 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.0 (3.94) | 42.0 (6.44) | 40.66 (6.74) | 43.33 (4.84) | 42.67 (5.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 20 | 20 | 20 | 20 | 80
Region of Enrollment [Number; unit: participants]
  Brazil | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: "Drinking Days" in the Previous Month
Description: The Alcohol Timeline Followback (TLFB) is a drinking assessment method that obtains estimates of daily drinking and has been evaluated with clinical and nonclinical populations. Using a calendar, people provide retrospective estimates of their daily drinking over a specified time period that can vary up to 12 months from the interview date.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Naltrexone | PUFAs | Naltrexone + PUFAs
Number analyzed (Participants) | 20 | 20 | 20 | 20
Days
  Number of "Drinking Days" Baseline | 19.54 (9.85) | 15.18 (10.32) | 17.75 (9.80) | 22.11 (11.63)
  Number of "Drinking Days" Final | 4.72 (8.74) | 5.66 (7.48) | 11.08 (12.87) | 11.12 (13.74)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone vs PUFAs vs Naltrexone + PUFAs; TIME COMPARISON; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Placebo vs Naltrexone vs PUFAs vs Naltrexone + PUFAs; GROUP COMPARISON; Test type: Superiority or Other; p = 0.69, ANOVA; Variance (F) = 0.71

2. Secondary Outcome: Short Alcohol Dependence Data Questionnaire (SADD)
Description: The Short Alcohol Dependence Data is a self-completion questionnaire designed to evaluate the presence and the degree of severity of alcohol dependence and consists of 15 questions. The minimum and maximum scores possible are 0 and 45 points respectively. The range of 1-9 is considered as low dependence, 10-19 medium dependence and 20 or more high dependence.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Naltrexone | PUFAs | Naltrexone + PUFAs
Number analyzed (Participants) | 20 | 20 | 20 | 20
Units on a Scale
  SADD Baseline | 34.90 (8.93) | 33.81 (9.92) | 31.91 (10.99) | 29.33 (11.11)
  SADD Final | 7.81 (11.93) | 11.36 (14.29) | 7.81 (11.93) | 9.16 (11.16)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone vs PUFAs vs Naltrexone + PUFAs; TIME COMPARISON; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Placebo vs Naltrexone vs PUFAs vs Naltrexone + PUFAs; GROUP COMPARISON; Test type: Superiority or Other; p = 0.53, ANOVA; Variance (F) = 0.73

3. Secondary Outcome: Obsessive Compulsive Drinking Scale (OCDS)
Description: The Obsessive Compulsive Drinking Scale (OCDS) is consisted by 14 items rated 0 - 4. The minimum and maximum values possibly obtained in this scale are respectively 0 and 56, this last one, meaning the most craving possible experienced. It is a short and easy to administer scale (average of 5 minutes per self-rating), built to measure severity and improvement during alcoholism treatment trials.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Naltrexone | PUFAs | Naltrexone + PUFAs
Number analyzed (Participants) | 20 | 20 | 20 | 20
Units on a Scale
  OCDS Baseline | 45.36 (9.86) | 42.45 (12.56) | 36.5 (14.88) | 37.55 (10.47)
  OCDS Final | 13.18 (14.98) | 11.81 (15.09) | 19.16 (20.93) | 14.00 (13.70)
Statistical Analysis 1: Comparison: Placebo vs Naltrexone vs PUFAs vs Naltrexone + PUFAs; TIME COMPARISON; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Placebo vs Naltrexone vs PUFAs vs Naltrexone + PUFAs; GROUP COMPARISON; Test type: Superiority or Other; p = 0.37, ANOVA; Variance (F) = 1.08

ADVERSE EVENTS:
Arm/Group | Placebo | Naltrexone | PUFAs | Naltrexone + PUFAs
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 1/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Naltrexone (N=20) | PUFAs (N=20) | Naltrexone + PUFAs (N=20)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No